CLINICAL TRIAL: NCT06668623
Title: Effect of Reiki on Neuropathic Pain Severity and Sleep Quality in Patients With Diabetic Neuropathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Fatma Gonul Burkev, Principal Investigator, Kayseri City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2024-SBB-0784; 76397871 (Other: Kayseri City Hospital)
Record Dates: First submitted 2024-10-26; First posted 2024-10-31 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Diabetic Neuropathy
Keywords: Diabetic Neuropathy; Pain; Sleep Quality; Reiki
MeSH Terms: conditions — Diabetic Neuropathies; Pain; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Reiki Group (Active Comparator): Remote Reiki application will be performed once a day for 20 minutes for four days by a researcher who has received second-level training.
  Interventions: Other: Reiki Group
- Sham Reiki Group (Sham Comparator): In the placebo group, the Sham Reiki group will receive remote Reiki application in accordance with the application protocol by a nurse who is not a Reiki practitioner trained by the researcher and has not received any previous training.
  Interventions: Other: Sham Reiki Group
- control group (No Intervention): For four weeks, patients will not receive any treatment. Individuals will continue to receive their normal treatments.

INTERVENTIONS:
Other: Reiki Group — Remote Reiki application will be performed once a day for 20 minutes for four days by a researcher who has received second level training. No changes will be made to the standard treatment plan of the patients during the application.
  Arms: Reiki Group
Other: Sham Reiki Group — In the placebo group, the Sham Reiki group will receive remote Reiki application in accordance with the application protocol by a nurse who is not a Reiki practitioner trained by the researcher and has not received any previous training.
  Arms: Sham Reiki Group

SUMMARY:
The study is planned to be conducted in a mixed research design with quantitative and qualitative types. The quantitative phase of the study was planned as a single-blind, randomized controlled study with Reiki group, Sham Reiki group and control group designs in order to examine the effect of second-level (remote application) Reiki applied to patients with diabetic neuropathy for 20 minutes a day for four days on pain intensity, neuropathic pain intensity (DN4 Questionnaire) total scores and sleep quality. The qualitative study will be conducted with 4 people from the Reiki and Sham Reiki groups, a total of 8 patients, one week after the application, using the individual in-depth interview method and a semi-structured questionnaire.

DETAILED DESCRIPTION:
Research hypotheses;

H01: Second-level Reiki applied to patients with diabetic neuropathy for 20 minutes once a day for 4 days has no effect on reducing pain intensity.

H11: Second-level Reiki applied to patients with diabetic neuropathy for 20 minutes once a day for 4 days has an effect on reducing pain intensity.

H02: Second-level Reiki applied to patients with diabetic neuropathy for 20 minutes once a day for 4 days has no effect on reducing neuropathic pain intensity.

H12: Second-level Reiki applied to patients with diabetic neuropathy for 20 minutes once a day for 4 days has an effect on reducing neuropathic pain intensity.

H03: Second-level Reiki applied to patients with diabetic neuropathy for 20 minutes once a day for 4 days has no effect on sleep quality.

H13: Second-level Reiki applied to patients with diabetic neuropathy for 20 minutes once a day for 4 days has an effect on sleep quality.

Reiki/Sham Reiki Application Protocol After the assignment of patients with diabetic neuropathy to the groups by lot, the Reiki group will be applied remotely by a researcher who has received second-level training, and the Sham Reiki group will be applied remotely by a nurse who is not a Reiki practitioner trained by the researcher and has not received any training before, in accordance with the application protocol.

Research Groups Intervention Group-1 A 20-minute remote Reiki application will be applied once a day for four days by a researcher who has received second-level training. No changes will be made to the standard treatment plan of the patients during the application.

Intervention Group-2 A 20-minute remote Sham Reiki application will be applied once a day for four days by a nurse who has not received Reiki training and has not been initiated. No changes will be made to the standard treatment plan of the patients during the application.

Control Group No application will be applied to the patients for four weeks. Individuals will continue to receive their normal treatments.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* No communication problems
* Communicating in Turkish
* No diagnosis of mental illness
* Willingness to participate in the study
* Being competent enough to answer forms and surveys
* VAS pain intensity 3 and above
* 4 Question Neuropathic Pain score 4 and above
* Not having received Reiki treatment

Exclusion Criteria:

* Receiving a different illness and treatment during the therapy process
* Leaving Reiki practice
* Psychiatric illness
* Becoming a Reiki practitioner or instructor
* Cerebrovascular disease
* Receiving Reiki practice

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale(VAS) | Pre-test data will be collected before starting the study and post-test data will be collected 1 week later.
  The value of "0 points" in the scale, which indicates the absence of pain, indicates a good condition, and the maximum value, "10 points", indicates a bad condition with unbearable pain intensity.

SECONDARY OUTCOMES:
McGill Pain Scale - Short Form | Pre-test data will be collected before starting the study and post-test data will be collected 1 week later.
  The scale form provides information on the sensory intensity, size and perceived effects of pain. In this respect, the scale consists of three dimensions. The first dimension includes 15 items that define the quality of pain. 11 of the items are sensory and 4 determine the perceptual dimension of pain. The intensity of pain is indicated in the items by grading between 0-3 (0=none, 1=mild, 2=moderate, 3=excessive). In the first dimension, the perceptual pain score is evaluated between 0-12, the sensory pain score is evaluated between 0-33 and the total pain score is evaluated between 0-45. An increase in the total score indicates an increase in the pain level. In the second dimension, the intensity of pain felt by the individual is determined by five expressions ranging from "mild pain" to "unbearable pain". In the third dimension, the individual's instant intensity is compared visually.
  The scale is listed in 0-5 points options. Minimum ''0=point, no pain; Indicates good condition.

OTHER OUTCOMES:
4 Question Neuropathic Pain Questionnaire (DN4) | Pre-test data will be collected before starting the study and post-test data will be collected 1 week later.
  The first two questions are based on interviews with the patient; The first question is about the definition of pain (tingling, burning, cold), and the second question is; It is related to paresthesia and dysesthesia (numbness, prickling, tingling and itching) in the painful area. The third question examines sensory disturbances (needling, touch and hypoesthesia) in the area where the pain is localized, and the fourth question; It determines whether friction causes an increase in the presence and severity of pain.
  Each question is scored as "yes answer = 1 point" or "no answer = 0 point". A minimum score of 4 points and above indicates neuropathic pain. Indicates a bad situation.
  A maximum score of 10 is taken from the scale. This indicates that the pain is severe and worse.
Pittsburgh Uyku Kalitesi Endeksi PUKI | Pre-test data will be collected before starting the study and post-test data will be collected 1 week later.
  Each item is evaluated between 0-3 points. The scale consists of 7 subcomponents that evaluate objective sleep quality (component 1), sleep latency (component 2), sleep duration (component 3), sleep habits, sleep disorders, sleeping pill use (component 5, component 6) and loss of daytime functionality. The sum of these components is the PSQI score. It indicates that sleep disturbance is severe in at least two of the 7 components or moderate in three component areas. A minimum score of 0-5 on the scale indicates that sleep quality is good. 5 points and above indicate that sleep quality is poor.
  Maximum scale total score It is 21 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Kayseri City Hospital, Kayseri, Kocasinan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Once the study is completed, its results will be shared with other researchers once the study data is published.